CLINICAL TRIAL: NCT04222192
Title: Evaluation of Different Type Ultrasound Guided Epidural Block Methods ; Paramedian Sagittal and Transverse Interlaminar View
Brief Title: Different Type Ultrasound Guided Epidural Block Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator ,Assoc. PhD. M.D., Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2011-KAEK-25 2019/12-09
Record Dates: First submitted 2020-01-04; First posted 2020-01-09 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Epidural Anesthesia; Ultrasound
MeSH Terms: interventions — Anesthesia, Epidural

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Epidural application (Sham Comparator): Epidural catheter insertions with conventional (anatomical landmarks use) method
  Interventions: Other: Epidural block
- Paramedian sagittal application (Active Comparator): Epidural catheter insertions with real time ultrasound guided Paramedian sagittal approach
  Interventions: Other: Epidural block
- Transverse Interlaminar application (Active Comparator): Epidural catheter insertions with real time ultrasound guided Transverse Interlaminar approach
  Interventions: Other: Epidural block

INTERVENTIONS:
Other: Epidural block — Epidural catheter insertions

SUMMARY:
The nerve blocks applied with ultrasonography are used for pain and operation after many operations today.

Applications with ultrasonography shorten the processing time, reduce the amount of local anesthetic used and lead to fewer complications.

However, the use of ultrasonography is not so common in neuraxial regional anesthesia applications. In the literature, epidural applications accompanied by ultrasonography were applied with different approaches.

DETAILED DESCRIPTION:
In this study the investigators will used the two different ultrasound -guided epidural block approach .

Paramedian sagittal oblique and Transverse interlaminar. The investigators will used this two technique in epidural catheter placement using the real-time ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were in the American Society of Anesthesiologists (ASA) I-III class
* Patients whom need medical epidural anesthesia
* Patients with consent to participate in the study

Exclusion Criteria:

* Patients with a known history of back surgery
* Bleeding diathesis disorder
* Allergy to local anesthetics
* Patient refusal

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Number of needle routing | 20 minutes
  number of needle redirects forming successful block
Epidural catheter placement time | 20 minutes
  time (minutes) until the epidural catheter is inserted

SECONDARY OUTCOMES:
Epidural igne visibility degree | 20 minutes
  4 = Excellent visibility, 3 = Medium visibility, 2 = Weak visibility 1 = No visibility using a 4-point Likert scale by the practitioner
Difficulty of catheter placement | 30 minutes
  Assessed by the Practitioner using a 10-point scale, 0: easiest, 10: hardest)
distance measurement of neuraxial structures | 30 minutes
  Anterior and posterior complex distance measured during epidural administration.
  Distance from skin to anterior aspect of ligament flavum (cm)
  Distance from skin to posterior dura (cm)
Patient position | 20 minutes
  Patient position during epidural placement Sitting Lateral

CONTACTS AND LOCATIONS:
Overall Officials: Korgün Ökmen, Assoc. PhD., Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Turkey (Türkiye)